CLINICAL TRIAL: NCT02487992
Title: The Randomized, Controlled, Multicenter Clinical Trial of CIK Plus S-1 and Bevacizumab as Maintenance Treatment for Patients With Advanced Colorectal Cancer
Brief Title: The Study of CIK Plus S-1 and Bevacizumab as Maintenance Treatment for Patients With Advanced Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZYY-CRC-001
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CIK plus S-1 and Bevacizumab (Experimental): Cytokine-Induced Killer Cells are used to treat advanced colorectal cancer patients with S-1 and Bevacizumab.
  S-1, 60mg,p.o.,Bid,d2-15. Bevacizumab (Avastin),7.5mg/kg,ivgtt,d1. 3 weeks is a cycle. Continue until the disease progress.
  Cytokine-induced killer cells 3 cycles,every 1 year. Continue until the disease progress.
  Interventions: Biological: Cytokine-Induced Killer Cells
- S-1 and Bevacizumab (No Intervention): S-1 is an oral anticancer agent, is a derivative of fluorouracil. Bevacizumab (Avastin) is a recombinant human monoclonal IgG1 antibody, which plays a role in the biological activity of human vascular endothelial growth factor. Bevacizumab is mainly used in the treatment of advanced colorectal cancer.
  S-1, 60mg,p.o.,Bid,d2-15. Bevacizumab (Avastin),7.5mg/kg,ivgtt,d1. 3 weeks is a cycle. Continue until the disease progress.

INTERVENTIONS:
Biological: Cytokine-Induced Killer Cells — CIK cells transfected with cytokine genes possess an improved proliferation rate and a higher cytotoxic activity as compared to regular CIK cells.
  Arms: CIK plus S-1 and Bevacizumab

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of cytokine-induced killer cell (CIK) plus S-1 and Bevacizumab vs S-1 and Bevacizumab as Maintenance Treatment for patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
1200 patients with stage Ⅳ colorectal cancer,who had received surgery and chemotherapy,will be randomly divided into group A（receive CIK plus S-1 and Bevacizumab ) or group B（just receive S-1 and Bevacizumab),and the randomize ratio will be 1:1. Patients in group A will receive 3 cycles of CIK treatment (every 1 year) and Apatinib (continuous).Patients in group B will receive only S-1 and Bevacizumab (continuous) .

ELIGIBILITY:
Inclusion Criteria:

* Patients who can accept curative operations 18-70 years old
* Histologically confirmed with colorectal cancer at stage Ⅳ
* Patients who can accept oral drugs;
* Eastern Cooperative Oncology Group (ECOG) performance status was 0 - 1.

Exclusion Criteria:

* Hemoglobin<8.0 g/dL,White blood cell <3 X 10^9/L;Platelet count <75 X 10^9/L; alanine aminotransferase, glutamic-oxalacetic transaminase, blood urine nitrogen and creatinine more than normal limits on 3.0 times
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Pregnant or lactating patients
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV) or TreponemaPallidun (TP) infection
* Patients who are suffering from serious autoimmune disease
* Patients who had used long time or are using immunosuppressant
* Patients who had active infection
* Patients who are suffering from serious organ dysfunction
* Patients who are suffering from other cancer
* Other situations that the researchers considered unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2015-07; Primary Completion 2043-07 (Estimated); Study Completion 2045-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | 3 months

SECONDARY OUTCOMES:
Disease-free survival | 3 months

OTHER OUTCOMES:
Adverse events | 1 months